CLINICAL TRIAL: NCT01306890
Title: A Registry of Sipuleucel-T Therapy in Men With Advanced Prostate Cancer
Acronym: PROCEED
Status: Completed | Type: Observational
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Other Study IDs: P10-3
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Advanced Prostate Cancer; Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sipuleucel-T
  Interventions: Biological: sipuleucel-T

INTERVENTIONS:
Biological: sipuleucel-T — Each dose of sipuleucel-T contains a minimum of 50 million autologous CD54+ cells activated with PAP-GM-CSF. The recommended course of therapy for sipuleucel-T is 3 complete doses, given at approximately 2-week intervals.
  Other Names: PROVENGE, APC8015

SUMMARY:
The purpose of this study is to further quantify the risk of cerebrovascular events (CVEs) following sipuleucel-T (PROVENGE®) therapy, and to follow all subjects for survival.

DETAILED DESCRIPTION:
Subjects will receive product as described in the sipuleucel-T approved label. The registry will be strictly observational and thus no additional clinical visits or laboratory tests will be conducted beyond normal clinical practice. Investigators will be asked to record information that becomes available in the normal course of clinical management.

ELIGIBILITY:
Inclusion Criteria:

* subjects must be at least 18 years of age
* subjects with advanced prostate cancer who will receive sipuleucel-T or who underwent their first leukapheresis for manufacture of sipuleucel-T ≤ 6 months prior to enrollment
* subjects must understand and sign an informed consent form

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men at least 18 years of age that have advanced prostate cancer that is treated with sipuleucel-T
Sampling Method: Non-Probability Sample
Enrollment: 1976 (Actual)
Dates: Start 2011-01-27 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Brown, MD, Study Director — Dendreon Pharmaceuticals
Locations (312):
- United States (312):
  - Birmingham Hematology and Oncology Associates, LLC, Bessemer, Alabama
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Ironwood Cancer and Research, Chandler, Arizona
  - Palo Verde Cancer Specialists, Glendale, Arizona
  - Weatern Regional Medical Center / Cancer Treatment Centers of America, Goodyear, Arizona
  - 21st Century Oncology, Scottsdale, Arizona
  - Pinnacle Oncology Hematology, Oncology Research Associates, PLLC, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - El Dorado Research, Tucson, Arizona
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - Little Rock Hematology Oncology: A Division of CARTI, Little Rock, Arkansas
  - South County Hematology/Oncology, Chula Vista, California
  - Wilshire Oncology Medical Group, Inc., Corona, California
  - Urology Specialists of Southern California, Encino, California
  - Robert A. Moss, M.D., F.A.C.P., Inc, Fountain Valley, California
  - Pacific Shores Medical Group, Glendale, California
  - Wilshire Oncology Medical Group, Inc., Glendora, California
  - Pacific Shores Medical Group, Huntington Beach, California
  - UCSD Medical Center - La Jolla, La Jolla, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Cancer Center Oncology Medical Group, La Mesa, California
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Pacific Shores Medical Group, Long Beach, California
  - Pacific Shores Medical Group, Los Alamitos, California
  - UCLA Institute of Urologic Oncology, UCLA Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Tower Urology, Los Angeles, California
  - Prostate Oncology Speciality Inc., Marina del Rey, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - North County Oncology Medical Group, Inc., Oceanside, California
  - Hematology-Oncology Medical Group of Orange County, Inc., Orange, California
  - Medical Oncology Care Associates (MOCA), Orange, California
  - The Center for Cancer Prevention and Treatment, St. Joseph Hospital, Orange, California
  - PMK Medical Group, Inc., DBA Ventura County Hematology Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical Group, Inc., Pasadena, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - Wilshire Oncology Medical Group, Inc., Rancho Cucamonga, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Cancer Center / Sacramento Center for Hematology and Medical Oncology, Sacramento, California
  - Sutter Memorial Hospital, Sacramento, California
  - UCSD Medical Center - Hillcrest, San Diego, California
  - Genesis Research, San Diego, California
  - Medical Oncology Associates, San Diego, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Edward Alexson, MD, Inc., Santa Ana, California
  - Stockton Hematology Oncology Medical Group, Stockton, California
  - Contra Costa Oncology, Walnut Creek, California
  - Wilshire Oncology Medical Group, Inc., West Covina, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Western Oncology/Hematology Associates, PC, Golden, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Advanced Urology, PC, Parker, Colorado
  - Rocky Mountain Cancer Centers, Parker, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Grove Hill Clinical Research, Grove Hill Medical Center, Urology Center of Grove Hill, New Britain, Connecticut
  - Yale Urology, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - The Stamford Hospital, Stamford, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Howard University Cancer Center & Howeard University Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center, Aventura, Florida
  - Manatee Medical Research Institute, LLC, Bradenton, Florida
  - 21st Century Oncology, Crestview, Florida
  - Integrated Community Oncology Network, Fleming Island, Florida
  - 21st Century Oncology, Fort Myers, Florida
  - Florida Cancer Specialists, PL, Hudson, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Watson Clinic LLP, Center for Cancer Care & Research, Clark & Daughtrey Medical Group, PA, Lakeland, Florida
  - Northwest Florida Hematology Oncology PA, Lynn Haven, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - 21st Century Oncology, Naples, Florida
  - Premier Oncology, Naples, Florida
  - Florida Cancer Specialists, PL, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Atlantic Urological Associates, Orange City, Florida
  - Integrated Community Oncology Network, Orange Park, Florida
  - Integrated Community Oncology Network, Palatka, Florida
  - Sacred Heart Medical Oncology Groupl, Pensacola, Florida
  - Integrated Community Oncology Network, Saint Augustine, Florida
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Georgia Cancer Specialists - Alpharetta, Alpharetta, Georgia
  - Georgia Cancer Specialists - Athens, Athens, Georgia
  - Georgia Cancer Specialists - Emory Midtown, Atlanta, Georgia
  - Midtown Urology, Atlanta, Georgia
  - Atlanta Hematology Oncology Associates, Atlanta, Georgia
  - Peachtree Hematology-Oncology Consultants, PC, Atlanta, Georgia
  - Piedmont West, Atlanta, Georgia
  - Emory University Hospital, The Emory Clinic, Winship Cancer Institute, Atlanta, Georgia
  - Georgia Urology, PA, Atlanta, Georgia
  - Augusta Oncology Associates, PC, Augusta, Georgia
  - Northwest Georgia Oncology Centers, P.C., Austell, Georgia
  - Northwest Georgia Oncology Centers, P.C., Carrollton, Georgia
  - Northwest Georgia Oncology Centers, P.C., Cartersville, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Georgia Cancer Specialists - Stemmer, Decatur, Georgia
  - Northwest Georgia Oncology Centers, P.C., Douglasville, Georgia
  - Gwinnett Hospital System Inc. dba Center for Cancer Care, Duluth, Georgia
  - Georgia Cancer Specialists - Fayetteville, Fayetteville, Georgia
  - Gwinnett Hospital System Inc. dba Center for Cancer Care, Lawrenceville, Georgia
  - Georgia Cancer Specialists - Macon, Macon, Georgia
  - Georgia Cancer Specialists - Kennestone, Marietta, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Urology Enterprises, Marietta, Georgia
  - Harbin Clinic, Rome, Georgia
  - Georgia Cancer Specialists - Northside, Sandy Springs, Georgia
  - Gwinnett Hospital System Inc. dba Center for Cancer Care, Snellville, Georgia
  - Georgia Cancer Specialists - Stockbridge, Stockbridge, Georgia
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Urological Surgeons of Illinois, Kankakee, Illinois
  - Oncology Specialists, S.C., Niles, Illinois
  - Mid-Illinois Hematology & Oncology Associates, LTD, Normal, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Urological Associates, Inc., Evansville, Indiana
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Metropolitan Urology Clinical Research, Jeffersonville, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology, P. C., Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, Michiana Hematology Oncology, P.C., South Bend, Indiana
  - Michiana Hematology Oncology, P. C., Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Physician's Clinic of Iowa, P.C., Cedar Rapids, Iowa
  - Heartland Oncology & Hematology, PLLC, Council Bluffs, Iowa
  - Kansas City Urology Care, Overland Park, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Wichita Urology Group P.A, Wichita, Kansas
  - Jewish Hospital & St. Mary's Healthcare, Louisville, Kentucky
  - Louisiana Oncology Associates, Crowley, Louisiana
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Louisiana Oncology Associates, New Iberia, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Louisiana Oncology Associates, Opelousas, Louisiana
  - Northwest Louisiana Oncology Associates Of Highland Clinic, Shreveport, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Myron I Murdock MD LLC, Greenbelt, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Steward Sr. Elizabeth's Medical Center of Boston Inc., Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Medical Center - Woodhaven, Brownstown, Michigan
  - Henry Ford Medical Center - Fairlane, Dearborn, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Karmanos Cancer Institute at Farmington Hills, Farmington Hills, Michigan
  - Lakeland Hospital, Niles, Michigan
  - Henry Ford Medical Center - Columbus Center, Novi, Michigan
  - Michgan Institute of Urology, PC, Saint Clair Shores, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Michigan Institute of Urology, PC, Troy, Michigan
  - Michigan Institute of Urology, PC, Utica, Michigan
  - Henry Ford Medical Center- West Bloomfield, West Bloomfield, Michigan
  - Minnesota Oncology Hematology, P.A., Burnsville, Minnesota
  - Minnesota Oncology Hematology, P.A., Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - Minnesota Oncology Hematology, P.A., Fridley, Minnesota
  - Minnesota Oncology Hematology, P.A., Maplewood, Minnesota
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - University Of Minnesota, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - Minnesota Oncology Hematology, P.A., Saint Paul, Minnesota
  - Adult and Pediatric Urology, Sartell, Minnesota
  - Minnesota Oncology Hematology, P.A., Woodbury, Minnesota
  - The Jones Clinic, PC, New Albany, Mississippi
  - Family Cancer Center Foundation, Inc., Oxford, Mississippi
  - Family Cancer Center Foundation, Inc., Southaven, Mississippi
  - St. Louis Cancer Care, LLP, Bridgeton, Missouri
  - St. Louis Cancer Care, LLP, Chesterfield, Missouri
  - Ellis Fischel Cancer Center - University of Missouri Health Care, Columbia, Missouri
  - Saint Luke's Cancer Institute, Saint Luke's Hospital, Kansas City, Missouri
  - St. Louis Cancer Care, LLP, St Louis, Missouri
  - Comprehensive Cancer Care, St Louis, Missouri
  - Nebraska Hematology-Oncology, PC, Lincoln, Nebraska
  - Southeast Nebraska Hematology & Oncology Consultants, PC / Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Urology Cancer Center & GU Research Network, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire
  - New Jersey Urology, LLC, Bloomfield, New Jersey
  - Oncology and Hematology Specialists, P.A., Denville, New Jersey
  - Hematology-Oncology Associates of Northern NJ, PA; Carol G. Simon Cancer Center, Morristown, New Jersey
  - Delaware Valley Urology, LLC, Mount Laurel, New Jersey
  - Sparta Cancer Center, Sparta, New Jersey
  - Urology Group of New Jersey, West Orange, New Jersey
  - New Mexico Oncology Hematology Consultants, LTD, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - The Jonah Center, Buffalo, New York
  - Zale P. Bernstein, MD, PC, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore Hematology/Oncology Associates, East Setauket, New York
  - Queens Medical Associates, Fresh Meadows, New York
  - NYU Clinical Cancer Center, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Integrated Medical Professionals, North Hills, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - Staten Island Urological Research, PC, Staten Island, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - Albert Einstein Cancer Center at the Montefiore Medical Park, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Asheville Hematology & Oncology, Asheville, North Carolina
  - Raleigh Hematology Oncology Associates, D.B.A., Cancer Centers of North Carolina, Cary, North Carolina
  - Presbyterian Hospital Cancer Center, Charlotte, North Carolina
  - Regional Cancer Care, P.A., Durham, North Carolina
  - Duke University Medical Center - Duke South Clinics, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Carolina Urology Partners, Gastonia, North Carolina
  - Presbyterian Hospital Huntersville, Huntersville, North Carolina
  - Matthews Hematology Oncology Associates, Matthews, North Carolina
  - Presbyterian Hospital Matthews, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists, Mooresville, North Carolina
  - Coastal Carolina Health Care, PA, dba New Bern Cancer Care, New Bern, North Carolina
  - Raleigh Hematology Oncology Associates, D.B.A., Cancer Centers of North Carolina, Raleigh, North Carolina
  - TriState Urologic Services PSC, Inc. dba TUG Research, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - SouthWest Urology, Middleburg Heights, Ohio
  - Cancer Centers of Southwest Oklahoma, Altus, Oklahoma
  - Cancer Centers of Southwest Oklahoma, Duncan, Oklahoma
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Urologic Specialists of Oklahoma, Tulsa, Oklahoma
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Providence Cancer Center Oncology and Hematology Care, Portland, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Urology Health Specialists, LLC, Bryn Mawr, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - UPMC Cancer Center / Hillman Cancer Centerl, Pittsburgh, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Center of Spartanburg, Spartanburg, South Carolina
  - Lexington Oncology Associates, LLC, West Columbia, South Carolina
  - Avera Cancer Institute, Avera Medical Group Oncology and Hematology, Sioux Falls, South Dakota
  - Family Cancer Center Foundation, Inc., Bartlett, Tennessee
  - The Jones Clinic, PC, Germantown, Tennessee
  - Family Cancer Center Foundation, Inc., Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Tennessee Oncology, Centennial Medical Center, Nashville, Tennessee
  - Urology Associates, P.C., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Hendrick Medical Center / Hendrick Cancer Center, Abilene, Texas
  - Texas Oncology-Abilene, Abilene, Texas
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncolocy - South Austin, Austin, Texas
  - Texas Oncology - Austin North, Austin, Texas
  - Texas Oncology - Beaumont, Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology - Cedar Park, Cedar Park, Texas
  - Cancer Specialists of South Texas, PA, Corpus Christi, Texas
  - Urology Clinics of North Texas, PLLC, Dallas, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Grandview, El Paso, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Gateway, El Paso, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Joe Battle, El Paso, Texas
  - Texas Oncology - Fort Worth 12th Avenue, Fort Worth, Texas
  - Texas Oncology - Southwest Fort Worth, Fort Worth, Texas
  - UTHealth Oncology, Memorial Hermann Cancer Center, Houston, Texas
  - Memorial Hennann Hosptial - Southwest Cancer Center, Houston, Texas
  - Memorial Hennann Hospital - Northeast Cancer Center, Humble, Texas
  - Texas Oncology - Kyle, Kyle, Texas
  - Texas Oncology - Lewisville, Lewisville, Texas
  - Texas Oncology - Seton-Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock, Round Rock, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Oncology San Antonio Research, LLC, San Antonio, Texas
  - Texas Oncology - San Marcos, San Marcos, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - Texas Oncology - Deke Slayton Cancer Center, Webster, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Urology of Virginia / SMG, Norfolk, Virginia
  - Harrison Poulsbo Hematology & Oncology, Poulsbo, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Medical Oncology Associates, PS, Spokane, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Wheaton Franciscan Healthcare - Elmbrook Memorial Hospital, Brookfield, Wisconsin
  - Wheaton Franciscan Healthcare - Reiman Cancer Center, Franklin, Wisconsin
  - Wheaton Franciscan Healthcare - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Wheaton Franciscan Healthcare - St. Francis Hospital, Milwaukee, Wisconsin
  - Wheaton Franciscan Healthcare -Wauwatosa Cancer Care, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Wei XX, Kwak L, Hamid A, He M, Sweeney C, Flanders SC, Harmon M, Choudhury AD. Outcomes in men with metastatic castration-resistant prostate cancer who received sipuleucel-T and no immediate subsequent therapy: experience at Dana Farber and in the PROCEED Registry. Prostate Cancer Prostatic Dis. 2022 Feb;25(2):314-319. doi: 10.1038/s41391-022-00493-x. Epub 2022 Feb 10. PMID 35145218
- [Derived] Sartor O, Armstrong AJ, Ahaghotu C, McLeod DG, Cooperberg MR, Penson DF, Kantoff PW, Vogelzang NJ, Hussain A, Pieczonka CM, Shore ND, Quinn DI, Small EJ, Heath EI, Tutrone RF, Schellhammer PF, Harmon M, Chang NN, Sheikh NA, Brown B, Freedland SJ, Higano CS. Survival of African-American and Caucasian men after sipuleucel-T immunotherapy: outcomes from the PROCEED registry. Prostate Cancer Prostatic Dis. 2020 Sep;23(3):517-526. doi: 10.1038/s41391-020-0213-7. Epub 2020 Feb 28. PMID 32111923

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sipuleucel-T
Started | 1976
Completed | 457 (Subjects were alive at the end of the study and had completed at least 3 years of follow up.)
Not Completed | 1519
Not completed — Adverse Event | 2
Not completed — Death | 1223
Not completed — Lost to Follow-up | 58
Not completed — Withdrawal by Subject | 88
Not completed — Unspecified reasons | 104
Not completed — Study Termination | 3
Not completed — No discontinuation documentation | 41

BASELINE CHARACTERISTICS:
Population: The analysis population only includes subjects that received at least one partial infusion of Sip-T.
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 1902
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 441
  >=65 years | 1461
Age, Continuous [Mean (Full Range); unit: Years] | 71.9 [42 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1902
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 221
  White | 1649
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1902
Weight [Mean (Standard Deviation); unit: kilogram] | 91.97 (17.67)
Height [Mean (Standard Deviation); unit: Centimeters] | 176.59 (7.29)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead
  Participants
    ECOG 0=Fully Active; No restrictions | 1265
    ECOG 1= Restricted Strenuous Activity | 571
    ECOG 2= Capable of selfcare | 34
    ECOG 3= Capable of limited selfcare | 8
    ECOG Not Reported | 24
Primary Gleason Score [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleason Score ≤3 | 486
    Gleason Score ≥4 | 1145
    Primary Gleason Score Data Not Recorded | 271
Gleason Sum Reported [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleason Score ≤7 | 790
    Gleason Score ≥8 | 963
    Gleson Sum Data Not Recorded | 149
Comorbidity Score [Count of Participants; unit: Participants] — The NCI Comorbidity Index was used for this study. It is a weighted index to predict risk of death within 1 year of hospitalization for patients with specific comorbid conditions. Nineteen conditions were included in the index. Each condition was assigned a weight from 1 to 6, based on the estimated 1-year mortality hazard ratio from a Cox proportional hazards model. These weights were summed and for this study, a score of 0-1 was classified as a LOW score and a score great than 2 was classified as a HIGH score.
  Participants
    High | 220
    Low | 1682
Alkaline phosphatase [Mean (Standard Deviation); unit: U/L] | 117.8 (163.2)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 12.68 (1.48)
Lactate dehydrogenase [Mean (Standard Deviation); unit: U/L] | 225.1 (211.6)
Prostate-specific antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 71.93 (287.89)

OUTCOME MEASURES:

1. Primary Outcome: To Further Quantify the Risk of Cerebrovascular Events Following Sipuleucel-T Therapy for All Subjects
Description: The incidence rate of CVEs (cardiovascular events) was estimated as the number of new events per 100 patient years of follow-up in the overall sample of men with advanced-stage or metastatic prostate cancer and in men with or without castration.
Time Frame: Every 3 months for a minimum of 3 years
Measure: Number; unit: events per 100 patient years
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 1902
events per 100 patient years | 1.2

2. Secondary Outcome: Survival
Description: To quantify survival by estimating the median time of survival in all subjects using the Kaplan-Meier method.
Time Frame: Every 3 months for a minimum of 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 1902
months | 30.7 [28.6 to 32.2]

ADVERSE EVENTS:
Time Frame: All SAEs reported or observed during or following the first infusion through 60 days post final infusion were recorded in subject's medical record and reported on an electronic case report form (eCRF). Data collection continued until every subject had been followed for minimum 3 years, had died, or had otherwise gone off study.
Arm/Group | Sipuleucel-T
All-Cause Mortality (participants affected / at risk) | 1223/1976
Serious Adverse Events (participants affected / at risk) | 260/1902
Other Adverse Events (participants affected / at risk) | 12/1902
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=1902)
Anaemia (Blood and lymphatic system disorders) | 7 (14)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (3)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (8)
Cardiac failure congestive (Cardiac disorders) | 4 (7)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 6 (7)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Papilloedema (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Intestinal ulcer (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (10)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (8)
Asthenia (General disorders) | 3 (6)
Chest pain (General disorders) | 6 (8)
Chills (General disorders) | 13 (18)
Death (General disorders) | 1 (2)
Disease progression (General disorders) | 28 (37)
Gait disturbance (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Pain (General disorders) | 1 (3)
Pyrexia (General disorders) | 6 (10)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Jaundice (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (2)
Device related infection (Infections and infestations) | 10 (10)
Device related sepsis (Infections and infestations) | 4 (4)
Endocarditis staphylococcal (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Intervertebral discitis (Infections and infestations) | 1 (1)
Ludwig angina (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (2)
Otitis media acute (Infections and infestations) | 1 (1)
Pneumococcal bacteraemia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (7)
Salmonella sepsis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (5)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (8)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (8)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 6 (13)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (2)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (11)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 2 (2)
Central nervous system haemorrhage (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 5 (6)
Cerebral infarction (Nervous system disorders) | 4 (5)
Cerebrovascular accident (Nervous system disorders) | 16 (20)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (2)
Haemorrhage intracranial (Nervous system disorders) | 4 (4)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hemiparesis (Nervous system disorders) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hydromyelia (Nervous system disorders) | 1 (1)
Intracranial mass (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Lacunar infarction (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 4 (4)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (3)
Syncope (Nervous system disorders) | 12 (12)
Thalamic infarction (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 6 (7)
Acute psychosis (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (5)
Depression (Psychiatric disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 8 (13)
Bladder obstruction (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (5)
Hydronephrosis (Renal and urinary disorders) | 1 (2)
Nephropathy (Renal and urinary disorders) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (3)
Renal injury (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (3)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Prostatomegaly (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fracture reduction (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Urethral stent insertion (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 8 (10)
Hot flush (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (5)
Ischaemia (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=1902)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (3)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No